CLINICAL TRIAL: NCT06764186
Title: A Phase IIIB Study to Evaluate the Use of Capivasertib in Combination With Fulvestrant in Patients With HR+ / HER2- Advanced Breast Cancer Who Have Relapsed/Progressed on ET and CDK4/6 Inhibitor Reflecting Real World Clinical Practice in Spain
Brief Title: A Phase IIIB Study to Evaluate the Use of Capivasertib in Combination With Fulvestrant in Patients With Advanced Breast Cancer Who Have Relapsed/Progressed on ET and CDK4/6 Inhibitor Reflecting Real World Clinical Practice in Spain
Acronym: CAPItana
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Apices Soluciones S.L. (Industry); SOLTI Breast Cancer Research Group (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D3612L00005
Record Dates: First submitted 2024-11-28; First posted 2025-01-08 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Locally Advanced or Metastatic Breast Cancer
Keywords: Luminal; PIK3CA/AKT1/PTEN; PI3K/AKT pathway; capivasertib; HR+ / HER2-; fulvestrant
MeSH Terms: conditions — Breast Neoplasms | interventions — Fulvestrant; capivasertib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Capivasertib + fulvestrant (Experimental): Fulvestrant: 2 intramuscular injections of 500 mg given on Day 1 of Weeks 1 and 3 of cycle 1, and then on Day 1, Week 1 of each cycle thereafter.
  Capivasertib: 400 mg (2 oral tablets) BD given on an intermittent weekly dosing schedule. Dosed on Days 1 to 4 in each week of a 28-day treatment cycle.
  Interventions: Drug: Fulvestrant; Drug: Capivasertib

INTERVENTIONS:
Drug: Fulvestrant — 2 intramuscular injections of 500 mg given on Day 1 of Weeks 1 and 3 of cycle 1, and then on Day 1, Week 1 of each cycle thereafter.
Drug: Capivasertib — 400 mg (2 oral tablets) BD given on an intermittent weekly dosing schedule. Dosed on Days 1 to 4 in each week of a 28-day treatment cycle

SUMMARY:
The purpose of this study is to evaluate the effectiveness and safety of capivasertib + fulvestrant treatment administration in patients with locally advanced (inoperable) or metastatic HR+ / HER2- breast cancer with PIK3CA/AKT1/PTEN-altered following recurrence or progression on or after endocrine therapy and CDK4/6 inhibitor.

DETAILED DESCRIPTION:
Phase IIIb, multicentre, single arm, Spain study assessing effectiveness/safety of capivasertib+fulvestrant in locally advanced (inoperable) or metastatic HR+/HER2- BC with the PIK3CA/AKT1/PTEN-altered following recurrence or progression on or after endocrine therapy and CDK4/6 inhibitor. Capivasertib will be administered as 400mg BD, 4 days on 3 days off in combination with fulvestrant at the approved dose of monthly 500mg (2 × 5mL IV), with an additional loading dose in Cycle 1.

ELIGIBILITY:
Key Inclusion Criteria

Histologically confirmed HR+/HER2- breast cancer (primary or metastatic):

* HR+ defined as ER+ with or without PRg+
* HER2- defined as IHC 0 or 1+, or IHC 2+/ISH-

Patient with tumours harbouring at least one PIK3CA/AKT1/PTEN qualifying alteration detected by a validated test (including NGS on tissue, cell block, or if tissue/cell block is not available, on ctDNA, as per protocol requirements. If alteration is initially detected by a method other than NGS, NGS on tissue/cell block must be performed within 45 days unless not available, which must be documented.)

Metastatic or locally advanced disease with radiological or objective evidence of recurrence or progression.

Patients must have received treatment with an ET in combination with CDK4/6i and have:

* Radiological evidence of breast cancer recurrence or progression while on, or within 12 months of the end of (neo)adjuvant treatment with an ET with CDK4/6i, OR
* Radiological evidence of progression while on prior ET with CDK4/6i administered as a treatment line for locally advanced or metastatic breast cancer.

Informed consent

Eastern Cooperative Oncology Group (ECOG)/ World Health Organisation (WHO) performance status ≤ 2 at enrollment (not more than 20% of patients with ECOG PS2 will be allowed).

Reproduction:

* Women of childbearing potential (WOCBP) patients with ovarian suppression induced by LHRH agonist should agree to use 2 forms of highly effective methods of accepted contraception to prevent pregnancy.
* Male patients should use barrier contraception.

Key Exclusion Criteria

History of another primary malignancy except for malignancy treated with curative intent with no known active disease ≥2 years before the first dose of study intervention and of low potential risk for recurrence.

Disease burden making the patient ineligible for endocrine therapy per the investigator judgement.

Unresolved toxicities from prior therapy greater than CTCAE grade 1.

Leptomeningeal metastases or symptomatic, unstable, or steroid-dependent brain metastases.

HbA1c ≥8.0% (63.9 mmol/mol).

Inadequate bone marrow reserve or organ function.

Severe or uncontrolled systemic diseases, uncontrolled hypertension, active infections including hepatitis B, hepatitis C, HIV, and confirmed COVID-19.

Known abnormalities in coagulation.

Refractory nausea, vomiting, malabsorption syndrome, chronic gastrointestinal diseases, inability to swallow formulated product, or significant bowel resection.

Previous allogenic bone marrow or solid organ transplant.

Known immunodeficiency syndrome.

Unknown or non-altered PIK3CA/AKT1/PTEN-status.

Evidence of dementia altered mental status or any psychiatric condition.

Pregnant women.

Participants with significant QT interval prolongation or a history of related cardiac conditions, including arrhythmias or recent cardiac procedures.

Prior/concomitant therapy:

* More than 2 lines of endocrine therapy or in combination with CDK4/6i for inoperable locally advanced or metastatic disease.
* More than 1 line of chemotherapy for inoperable locally advanced or metastatic disease. Adjuvant and neoadjuvant chemotherapy are not classed as lines of chemotherapy for ABC.

AKT1, PIK3CA and mTOR inhibitors not allowed.

Adequate washout or dose reduction may be required for some CYP3A.

Participation in another clinical study with a study intervention.

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2025-01-07 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Time to next treatment (TTNT) | From start of date of first dose of capivasertib+fulvestrant treatment to date of the first subsequent anti-cancer therapy or death or up to within approximately 12 months after Last Subject Inclusion
  Time to next treatment (TTNT1 is defined as the time from the date of first dose of capivasertib+fulvestrant until the first subsequent anti-cancer therapy after discontinuation of study treatment or death due to any cause).

SECONDARY OUTCOMES:
Number of patients with AEs. | From enrollment up to at least 30 days (+7 days) after last dose of capivasertib + fulvestrant treatment
  Safety and tolerability will be evaluated in terms of AEs, SAEs, and AESIs.
Time to first Subsequent Chemotherapy (TFSC) | From start of capivasertib+fulvestrant treatment to the first Subsequent Chemotherapy, death, withdrawal of consent or the end of study (approximately 24 months)
  TFSC is defined as the time from the date of first dose of capivasertib + fulvestrant treatment until the first date of the first cycle of the subsequent chemotherapy, or death from any cause.
Progression-free survival (PFS) | From date of first dose of Capivasertib + fulvestrant until date of disease progression, death, withdrawal of consent or the end of study (approximately 24 months)
  PFS is defined as time from the first dose of capivasertib + fulvestrant treatment to Response Evaluation Criteria in Solid Tumors (RECIST) 1.1-defined progressive disease as assess by the investigator or death due to any cause.
Objective Response Rate (ORR) | From start of capivasertib+fulvestrant treatment to progression/death or up to 6 months after Last Subject Inclusion
  Objective Response Rate (ORR) using site investigator assessments according to RECIST 1.1.
Overall survival (OS) | From date of first dose of capivasertib + fulvestrant treatment until death, withdrawal of consent, or the end of the study (approximately 24 months).
  OS is defined as the time from first dose of capivasertib + fulvestrant treatment until the date of death due to any cause.
Number of patients with change in EORTC QLQ C30 and QLQ-BR42, respectively | From start of capivasertib+fulvestrant treatment to first dose of subsequent line of treatment/death or up to within approximately 12 months after Last Subject Inclusion
  Change from baseline in score on EORTC QLQ-C30 and EORTC QLQ-BR42 reported at enrollment and then throughout the prospective study follow-up to end of the capivasertib + fulvestrant
Time to deterioration | From start of capivasertib+fulvestrant treatment to first dose of subsequent line of treatment/death or up to within approximately 12 months after Last Subject Inclusion
  Time to deterioration defined as the time from the date of the first dose of treatment until the date of the first clinically meaningful deterioration that is confirmed at a subsequent visit at least 14 days apart or death.
Number of patients with change from in PGI-S | From start of capivasertib+fulvestrant treatment to the end of the study (approximately 24 months)
  Change from baseline in score on the PGI-S to assess how a patient perceives the overall severity of cancer symptoms over the past 7 days at study enrollment and then weekly throughout the prospective study follow-up on study treatment
Number of patients with change in PGI-II | From start of capivasertib+fulvestrant treatment to the end of the study (approximately 24 months)
  Change from baseline in score on the PGI-TT to assess how a patient perceives the overall tolerability of the study treatment over the past 7 days at study enrollment and then weekly throughout the prospective study follow-up on study treatment
Number of patients with change in Daily bowel habits | From start of capivasertib+fulvestrant treatment to the end of the study (approximately 24 months)
  Change from baseline in score on the Daily bowel habits diary (BSFS) to classify the stools based on their appearance at study enrollment and then daily oughout the prospective study follow-up on study treatment
Number of patients with change in ADAQ | From start of capivasertib+fulvestrant treatment to the end of the study (approximately 24 months)
  Change from baseline in score on ADAQ to assess the adherence of capivasertib + fulvestrant treatment at study enrollment and then weekly throughout the prospective study follow-up on study treatment

CONTACTS AND LOCATIONS:
Locations (15):
- Spain (15):
  - Research Site, Alicante
  - Research Site, Barcelona
  - Research Site, Bilbao (Vizcaya)
  - Research Site, Córdoba
  - Research Site, Donostia / San Sebastian
  - Research Site, El Palmar
  - Research Site, Girona
  - Research Site, Madrid
  - Research Site, Oviedo
  - Research Site, Palma deMallorca
  - Research Site, Salamanca
  - Research Site, Santander
  - Research Site, Seville
  - Research Site, Valencia
  - Research Site, Zaragoza

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA PhRMA Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org.
  Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/